CLINICAL TRIAL: NCT03446495
Title: A Non-interventional, Multicenter Study of the Combination of Pegylated Liposomal Doxorubicin and Trabectedin in Routine Practice in Patients With Recurrent Partial-platinum Sensitive Ovarian Cancer
Brief Title: An Observational Study of Combination of Pegylated Liposomal Doxorubicin and Trabectedin in Routine Practice in Patients With Recurrent Partial-platinum Sensitive Ovarian Cancer
Acronym: Renaissance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Suriya Yessentayeva (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor-Investigator, Suriya Yessentayeva, Chair, Scientific Medical Society, Kazakhstan
Organization: Scientific Medical Society, Kazakhstan (Other)
Other Study IDs: R279741OVC4001
Record Dates: First submitted 2018-02-13; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer, trabectedin, recurrent ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Trabectedin; 1-dodecylpyridoxal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trabectedin + PLD: Trabectedin + PLD according to SmPC
  Interventions: Drug: Trabectedin + PLD

INTERVENTIONS:
Drug: Trabectedin + PLD — Combination of Trabectedin + PLD: PLD 30 mg/m2 intravenous (IV) infusion over 90 minutes + trabectedin 1.1 mg/m2 IV infusion over 3 hours every 3 weeks.

SUMMARY:
This is a Non-interventional, Multicenter study evaluating the efficacy and safety of the combination of pegylated liposomal doxorubicin and trabectedin in routine practice in patients with recurrent partial-platinum sensitive ovarian cancer, which is held in Kazakhstan.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Histologically proven epithelial ovarian cancer
* ECOG 0-1
* Partially platinum sensitive relapsed ovarian cancer: platinum-free interval 6 -12 months
* With 1-2 or more cycles on trabectedin treatment at the recommended dose of 1.1mg/m2 q3w 3hr infusion in combination of PLD at 30mg/ml with appropriate pre-medication
* Prior treatment with 1 or more chemotherapy regimen

Exclusion Criteria:

* Platinum resistant disease: PFI < 6 months (progression within six months after first-line platinum-based chemotherapy)
* Unwilling or unable to have a central venous catheter
* Patients with hepatic impairment (Patients with elevated bilirubin)
* Patients with renal impairment (Patients with serum creatinine >1.5 mg/dL)
* Patients with hematologic impairment (baseline neutrophil counts of less than 1,500 cells/mm3 and platelets count of less than 100,000 cells/mm3)
* Patients with serious impaired cardiac function (patients with cardiac disease and with reduction of the QRS complex)
* AIDS-related Kaposi's sarcoma
* Lactation or pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-03-20 (Estimated); Study Completion 2019-05-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Patient will be followed during 37 weeks
  ORR will be evaluated by Response Evaluation Criteria In Solid Tumors (RECIST V 1.1).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Patient will be followed during 37 weeks
  PFS is defined as the time from the 1st treatment cycle until objective tumor progression or death
Safety according to CTCAE v4.0 | Patient will be followed during 37 weeks
  To assess patient safety and the tolerance of trabectedin + PLD

CONTACTS AND LOCATIONS:
Locations (9):
- Kazakhstan (9):
  - Almaty oncological center, Almaty
  - Almaty regional oncological dispensary, Almaty
  - Kazakh institute of oncology and radiology, Almaty
  - Astana Oncology Center, Astana
  - Kyzylorda regional Oncological center, Kyzylorda
  - West Kazakhstan regional oncology dispensary, Oral
  - North Kazakhstan Regional Oncology Center, Petropavl
  - South Kazakhstan regional oncologic dispensary, Shymkent
  - East Kazakhstan Regional Oncology Dispensary, Ust-Kamenogorsk

IPD SHARING:
Plan to Share IPD: No